CLINICAL TRIAL: NCT00824902
Title: A Pilot Trial Evaluation of Ultrasound Elasticity/Tissue Strain-Hardening Imaging for Prostate Cancer in Patients Undergoing Radical Prostatectomy
Brief Title: Evaluation Ultrasound Elasticity/Tissue Strain-Hardening Imaging for Prostate Cancer Patients Undergoing Radical Prostatectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical Issues
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0949
Record Dates: First submitted 2009-01-15; First posted 2009-01-19 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2013-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostate; Radical Prostatectomy; Tissue Elastography; Tissue Elastography Imaging; Software Program Measuring Prostate Elasticity; Elasticity/Tissue Strain-Hardening Imaging; Ultrasound
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tissue Elastography Imaging (Experimental): Using special elastography software, probe pressed gently against prostate during routine ultrasound before prostate surgery, 10-15 minutes process.
  Interventions: Procedure: Tissue Elastography Imaging

INTERVENTIONS:
Procedure: Tissue Elastography Imaging — Using special elastography software, probe pressed gently against prostate during routine ultrasound before prostate surgery, 10-15 minutes process.

SUMMARY:
The primary objective is to perform a pilot trial evaluation of a novel prostate ultrasound imaging software utilizing tissue elasticity measurements to identify tumor foci among men who will undergo radical prostatectomy for localized prostate cancer.

As a secondary objective, investigators will compare elasticity measured tumor foci volume to the measured volume from radical prostatectomy pathologic examination.

DETAILED DESCRIPTION:
Study Imaging:

As part of routine care, ultrasound scanning is commonly used to find the cancerous areas of the prostate before the prostate is surgically removed. The ultrasound images are in black, white, and gray, and the dark areas may show prostate cancer.

In this study, standard ultrasound scanning will still be done, but researchers want to test another form of diagnostic imaging called tissue elastography.

Tissue elastography uses the same machine and probe as the ultrasound. The probe is gently pushed through the rectum and into the prostate gland (similar to a digital rectal exam). The ultrasound machine will use a special elastography software that is designed to scan the prostate for differences in how hard the tissue is. Prostate cancer tissue may be harder than surrounding tissue, and the images produced by tissue elastography are designed to show these differences in hardness of tissue.

Screening:

Before you can join this study, the study staff will review the results of your most recent prostate ultrasound and biopsy. This is a "screening" procedure to help the doctor decide if you are eligible to take part in this study.

Study Procedures:

If you are found to be eligible to take part in this study, tissue elastography imaging will be performed during your routine ultrasound before prostate surgery. The probe, once inserted, will be gently pressed against the prostate a few times in order to perform the tissue elastography. The routine ultrasound part of the procedure should take about 10 minutes, and the elastography should take about 10-15 minutes.

Length of Study Participation:

Your active participation in this study will be over after the tissue elastography imaging. The routine ultrasound will be the main decision-making exam. However, if the tissue elastography imaging shows something different and possibly related to your care, your doctor will be informed.

After the prostate is removed and the tissue results are available, researchers will compare the tissue results with the tissue elastography images. You will not receive the results of the tissue elastography imaging, as the imaging is being used for research only.

This is an investigational study. The ultrasound machine and probe that are used for the tissue elastography in this study are FDA approved for ultrasound scanning. Performing tissue elastography for prostate cancer detection is investigational. At this time and for this purpose, tissue elastography is only being performed in research.

Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients selected for radical prostatectomy (any technique) at MDACC
2. Histologic diagnosis of prostate cancer, clinical stage cT1c-cT3b
3. Serum prostate specific antigen less than 30 ng/ml.
4. Any Gleason score
5. Total prostate volume of 20-60 cc, measured by outside ultrasound or clinical examination at MDACC.
6. Group 1: high volume disease. At least 3 positive cores containing cancer on one side of the prostate Group 2: low volume disease. Less than 50% tumor length in a single positive core on one side of the prostate

Exclusion Criteria:

1. Prior radiation therapy to the pelvis
2. Prior hormonal therapy within 3 months (including LH/RH agonists, estrogens, testosterone receptor blockade, finasteride, dutasteride)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of diagnostic technique (using tissue elastography) for prostate cancer detection in men scheduled to undergo a radical prostatectomy | 2 Years
  Pilot evaluation of novel prostate ultrasound imaging software utilizing tissue elasticity measurements to identify tumor foci among men who will undergo radical prostatectomy for localized prostate cancer. The methods of Bland and Altman (1986) used to assess whether the tumor volume estimated by the ultrasound imaging technique agrees with the tumor volume measured at pathology. An ultrasound based elasticity measurement technique will detect differences in prostate hardness by using sophisticated mathematical techniques to analyze ultrasound images obtained before and after small compressions of the prostate gland with the ultrasound probe, detecting differences in hardness by measuring relative displacements of portions of the gland. Elasticity images obtained during standard, medically-indicated prostate sonography.

CONTACTS AND LOCATIONS:
Overall Officials: John W. Davis, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org